CLINICAL TRIAL: NCT07240701
Title: A Prospective, Single-Center, Randomized Controlled Trial Comparing Normal Saline and Ringer's Lactate for Initial Fluid Resuscitation in Adult Patients With Sepsis in the Emergency Department
Brief Title: Normal Saline Versus Ringer's Lactate for Initial Fluid Resuscitation in Sepsis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Egemen Yildiz (Other)
Responsible Party: Sponsor-Investigator, Egemen Yildiz, MD, Kutahya City Hospital
Organization: Kutahya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25-AKD-210
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Sepsis
Keywords: sepsis; Fluid Therapy; Saline Solution; Ringer's Lactate; Randomized Controlled Trial; Mortality; emergency department; Vasoconstrictor Agents; Renal Replacement Therapy; Crystalloid Solutions
MeSH Terms: conditions — Sepsis; Emergencies | interventions — Ringer's Lactate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two parallel groups receive either Ringer's lactate or 0.9% sodium chloride (normal saline) for initial fluid resuscitation in sepsis, with double-blind randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringer's Lactate Group (Experimental): Eligible participants in this group will receive Ringer's lactate solution as the initial intravenous fluid for resuscitating sepsis. This will be administered through a peripheral intravenous line at a rate of 1000 ml over 30-60 minutes, as determined by the attending physician and the patient's clinical condition. All other treatments will follow standard sepsis care protocols.
  Interventions: Other: Ringer's Lactate
- Normal Saline Group (Active Comparator): Eligible participants in this arm will receive 0.9% sodium chloride (normal saline) as the initial intravenous fluid for resuscitation in sepsis. This will be administered through a peripheral intravenous line at a rate of 1000 ml over 30-60 minutes, as determined by the attending physician and the patient's clinical condition. All other treatments will follow standard sepsis care protocols.
  Interventions: Other: Normal Saline (0.9% Sodium Chloride)

INTERVENTIONS:
Other: Ringer's Lactate — Intravenous infusion of Ringer's lactate solution for initial fluid resuscitation in sepsis. Each participant receives approximately 1000 mL of Ringer's lactate administered via a peripheral intravenous line over 30 to 60 minutes during the initial resuscitation phase. The intervention is performed once, and all subsequent management follows standard sepsis treatment protocols.
  Arms: Ringer's Lactate Group
Other: Normal Saline (0.9% Sodium Chloride) — Intravenous infusion of 0.9% sodium chloride solution (normal saline) for initial fluid resuscitation in sepsis. Each participant receives approximately 1000 mL of normal saline administered via a peripheral intravenous line over 30 to 60 minutes during the initial resuscitation phase. The intervention is performed once, and all subsequent management follows standard sepsis treatment protocols.
  Arms: Normal Saline Group

SUMMARY:
This clinical trial aims to determine if the type of intravenous fluid used for initial resuscitation affects the short-term outcomes of adult patients with sepsis who are treated in the emergency department.

The main questions it aims to answer are:

Does using Ringer's lactate instead of 0.9% sodium chloride (normal saline) reduce 24-hour mortality in patients with sepsis?

Does the type of fluid influence other short-term outcomes, such as the need for vasopressors, mechanical ventilation, hemodialysis, and length of hospital stay?

Researchers will compare two groups of participants:

* The Ringer's lactate group (intervention group)
* The 0.9% sodium chloride group (control group).

Participants will:

* Receive either Ringer's lactate or normal saline for initial fluid resuscitation as part of standard sepsis care.
* They will be observed for 24 hours to assess survival and other early outcomes.

DETAILED DESCRIPTION:
This prospective, single-center, randomized, double-blind, controlled clinical trial aims to compare the effects of Ringer's lactate and 0.9% sodium chloride (normal saline) solutions for initial fluid resuscitation in adult patients with sepsis who are treated in the emergency department. The study is conducted in accordance with the Surviving Sepsis Campaign's 2021 guidelines, which emphasize the importance of early and adequate crystalloid resuscitation in sepsis management. Although both solutions are widely used in clinical practice, evidence regarding their comparative effects on short-term mortality and organ dysfunction is inconsistent. This study seeks to provide prospective, blinded data to clarify whether fluid type influences early outcomes in patients with sepsis.

Participants who meet eligibility criteria will be randomized in a 1:1 ratio using a computer-generated sequence prepared by an independent staff member. To ensure blinding, study fluids will be provided in identical coded containers, and patients, treating clinicians, and investigators will remain unaware of the assigned fluid type throughout the study period.

The assigned study fluid will be administered intravenously as an initial bolus according to clinical judgment. After completion of the initial bolus, all subsequent fluid therapy and additional treatments will follow standard institutional practice at the discretion of the treating physician.

If clinical circumstances require breaking the study blind for patient safety reasons, the investigator will document the reason and unblind the allocation. There will be no delay in clinical management as a result of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients (≥18 years of age) presenting to the emergency department.
* Diagnosed or suspected sepsis secondary to an infectious cause.
* Provision of written informed consent by the patient, or if the patient is unable to consent, by a first-degree relative or legally authorized representative.

Exclusion Criteria:

* Age under 18 years old.
* Pregnant women.
* Informed consent was not obtained from the patient or their first-degree relative/legal guardian.
* Patients who are receiving cardiopulmonary resuscitation (CPR) or who require endotracheal intubation at the time of presentation.
* Patients with severe volume depletion unrelated to sepsis (e.g., diabetic ketoacidosis, burns, or active gastrointestinal bleeding).
* Patients with severe hyperkalemia (serum potassium level of at least 6.5 mmol/L with ECG changes).
* Patients with hypotension that is not related to sepsis (e.g., active hemorrhage or intracranial bleeding).
* Patients with clinical signs of pulmonary edema or congestive heart failure.
* Cases in which the treating physician determines that one isotonic crystalloid (Ringer's lactate or 0.9% NaCl) is clearly superior to the other due to clinical condition or comorbidities.
* Cases in which the treating physician anticipates that fluid therapy might be delayed due to study participation.
* Patients requiring immediate hospital or ICU admission before completion of initial emergency department resuscitation.
* Patients with sepsis sources requiring urgent invasive intervention known to directly affect mortality (e.g., an undrainable abscess or osteomyelitis).

Additional exclusion criteria based on the contraindications listed in the Ringer's lactate product information:,

* Known hypersensitivity to sodium lactate.
* Extracellular hyperhydration or hypervolemia.
* Severe renal failure with oliguria or anuria.
* Decompensated heart failure.
* Hypercalcemia.
* Metabolic alkalosis or severe metabolic acidosis.
* Conditions associated with impaired lactate metabolism, such as lactic acidosis, severe liver failure, and cirrhosis with ascites.
* Current use of digitalis preparations (e.g., digoxin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
24-hour All-Cause Mortality | Within 24 hours after initiation of fluid resuscitation
  The proportion of participants who die from any cause within 24 hours after receiving the assigned study fluid (Ringer's lactate or normal saline) for initial resuscitation. Mortality will be determined based on hospital medical records.

SECONDARY OUTCOMES:
Requirement for Vasopressor Support | Within 6 hours after initiation of fluid resuscitation
  The proportion of participants who receive any vasopressor agents (e.g. norepinephrine, epinephrine or vasopressin) within six hours of initial fluid administration, as documented in the medical record. Will be reported as a percentage.
Requirement for Mechanical Ventilation | Within 6 hours after initiation of fluid resuscitation
  The proportion of participants who require endotracheal intubation and mechanical ventilation within six hours of the initial administration of fluids. Will be reported as a percentage.
Requirement for Emergency Hemodialysis | Within 6 hours after initiation of fluid resuscitation
  The proportion of participants who require emergency hemodialysis within 6 hours after initial fluid administration. The outcome will be reported as a percentage.
Urine Output Response to Fluid Resuscitation | Within 6 hours after initiation of fluid resuscitation
  The proportion of participants with a total urine output of ≥3 mL/kg during the first six hours after receiving the study fluid, as recorded in the patient's follow-up chart. The outcome will be reported as a percentage.
Change in Serum Lactate Level | Baseline and 3 hours after initiation of fluid resuscitation
  Change in serum lactate concentration (mmol/L), calculated as the difference between the value at 3 hours and the baseline value obtained before fluid administration. The outcome will be reported as the mean change (mmol/L).
Length of Stay in Intensive Care Unit (ICU) | From ICU admission until ICU discharge, assessed up to 30 days
  Duration of ICU stay, measured in days among participants admitted to the ICU after initial fluid resuscitation.
Total Length of Hospital Stay | From hospital admission until hospital discharge, assessed up to 30 days
  Total duration of hospitalization, measured in days based on hospital records.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya City Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the study results will be shared upon reasonable request after publication. Shared data will include demographic, treatment, and outcome variables. Access will be granted to qualified researchers with ethics committee approval and a sound research proposal.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the main results and will remain available for 5 years thereafter. Requests received after this period will be evaluated on a case-by-case basis.
Access Criteria: Data will be shared with qualified researchers upon reasonable request. Interested investigators must submit a brief research proposal describing study aims, statistical analysis plan, and data protection procedures. Access will be granted after approval by the institutional ethics committee. The de-identified dataset and relevant documents will be shared electronically via a secure data transfer platform.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691